CLINICAL TRIAL: NCT01977612
Title: Randomized Controlled Phase IIB Trial Evaluating Wound Complication Rate After Skin Closure With Staples Versus Subcuticular Suture in Patients With BMI >=30
Brief Title: Randomized Clinical Trial of Skin Closure With Staples Versus Suture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201304058
Record Dates: First submitted 2013-04-17; First posted 2013-11-06 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Wound Infection; Wound Complication
Keywords: Wound infection; Wound separation; Skin staples; Subcuticular suture
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stainless Steel Staples (Active Comparator): Skin closure with stainless steel staples
  Interventions: Device: Stainless steel staples
- 4-0 monofilament Sutures (Experimental): Skin closure with 4-0 monofilament sutures
  Interventions: Device: 4-0 monofilament suture

INTERVENTIONS:
Device: 4-0 monofilament suture — Skin closure using 4-0 monofilament suture
  Other Names: 4-0 Monocryl suture
  Arms: 4-0 monofilament Sutures
Device: Stainless steel staples — Skin closure using stainless steel staples.
  Arms: Stainless Steel Staples

SUMMARY:
Women with gynecologic cancers are often obese and have other risk factors for post-operative wound separation. Data from obstetrics and orthopedic surgery literature have shown a decreased risk of wound separation and complications when the skin is closed with suture as compared to staples. Skin closure with either staples or suture is considered standard of care. Traditionally, most wounds have been closed with staples given their ease of use and quick application. In this randomized study the investigators plan to evaluate and compare the complication rate associated with both standard closures.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial to evaluate for a difference in wound complication rate between closure with sutures that are placed just below the skin level to hold the skin together and metal staples in obese women (BMI>=30) undergoing gynecologic or gynecologic oncology via a midline skin incision for benign or cancer indications under the supervision of one of the full-time faculty members of the Division of Gynecologic Oncology at Washington University School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* All women, >=18 and <= 85 years of age, undergoing surgery, via a midline laparotomy.
* Body mass index >=30
* Benign or oncologic indications for surgery.
* Women of childbearing age will be required to have a negative human chorionic gonadotropin (HCG) test within seven days of surgery.
* Surgery will be supervised by one of the gynecologic oncology attendings at Washington University School of Medicine.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Pfannenstiel or transverse abdominal incision
* Concomitant panniculectomy or plastic surgery
* Women <18 years of age
* History of prior abdominal or pelvic radiation
* Inability to sign an informed consent form prior to registration on study
* Inability to understand spoken or written English
* Prisoner
* Mental incapacity
* A history of allergic reactions attributed to either Monocryl suture or stainless steel staples.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Kuroki, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perencevich EN, Sands KE, Cosgrove SE, Guadagnoli E, Meara E, Platt R. Health and economic impact of surgical site infections diagnosed after hospital discharge. Emerg Infect Dis. 2003 Feb;9(2):196-203. doi: 10.3201/eid0902.020232. PMID 12603990
- [Background] Nugent EK, Hoff JT, Gao F, Massad LS, Case A, Zighelboim I, Mutch DG, Thaker PH. Wound complications after gynecologic cancer surgery. Gynecol Oncol. 2011 May 1;121(2):347-52. doi: 10.1016/j.ygyno.2011.01.026. Epub 2011 Feb 15. PMID 21324517
- [Background] Cardosi RJ, Drake J, Holmes S, Tebes SJ, Hoffman MS, Fiorica JV, Roberts WS, Grendys EC Jr. Subcutaneous management of vertical incisions with 3 or more centimeters of subcutaneous fat. Am J Obstet Gynecol. 2006 Aug;195(2):607-14; discussion 614-6. doi: 10.1016/j.ajog.2006.04.013. Epub 2006 Jun 21. PMID 16796988
- [Background] Gallup DC, Gallup DG, Nolan TE, Smith RP, Messing MF, Kline KL. Use of a subcutaneous closed drainage system and antibiotics in obese gynecologic patients. Am J Obstet Gynecol. 1996 Aug;175(2):358-61; discussion 362. doi: 10.1016/s0002-9378(96)70146-1. PMID 8765253
- [Background] Soisson AP, Olt G, Soper JT, Berchuck A, Rodriguez G, Clarke-Pearson DL. Prevention of superficial wound separation with subcutaneous retention sutures. Gynecol Oncol. 1993 Dec;51(3):330-4. doi: 10.1006/gyno.1993.1299. PMID 8112641
- [Background] Anthony T, Murray BW, Sum-Ping JT, Lenkovsky F, Vornik VD, Parker BJ, McFarlin JE, Hartless K, Huerta S. Evaluating an evidence-based bundle for preventing surgical site infection: a randomized trial. Arch Surg. 2011 Mar;146(3):263-9. doi: 10.1001/archsurg.2010.249. Epub 2010 Nov 15. PMID 21079110
- [Background] Magann EF, Chauhan SP, Rodts-Palenik S, Bufkin L, Martin JN Jr, Morrison JC. Subcutaneous stitch closure versus subcutaneous drain to prevent wound disruption after cesarean delivery: a randomized clinical trial. Am J Obstet Gynecol. 2002 Jun;186(6):1119-23. doi: 10.1067/mob.2002.123823. PMID 12066083
- [Background] Ramsey PS, White AM, Guinn DA, Lu GC, Ramin SM, Davies JK, Neely CL, Newby C, Fonseca L, Case AS, Kaslow RA, Kirby RS, Rouse DJ, Hauth JC. Subcutaneous tissue reapproximation, alone or in combination with drain, in obese women undergoing cesarean delivery. Obstet Gynecol. 2005 May;105(5 Pt 1):967-73. doi: 10.1097/01.AOG.0000158866.68311.d1. PMID 15863532
- [Background] Figueroa D, Jauk VC, Szychowski JM, Garner R, Biggio JR, Andrews WW, Hauth J, Tita AT. Surgical staples compared with subcuticular suture for skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Jan;121(1):33-8. doi: 10.1097/aog.0b013e31827a072c. PMID 23262925
- [Background] Frishman GN, Schwartz T, Hogan JW. Closure of Pfannenstiel skin incisions. Staples vs. subcuticular suture. J Reprod Med. 1997 Oct;42(10):627-30. PMID 9350017
- [Background] Cromi A, Ghezzi F, Gottardi A, Cherubino M, Uccella S, Valdatta L. Cosmetic outcomes of various skin closure methods following cesarean delivery: a randomized trial. Am J Obstet Gynecol. 2010 Jul;203(1):36.e1-8. doi: 10.1016/j.ajog.2010.02.001. Epub 2010 Apr 24. PMID 20417924
- [Background] de Graaf IM, Oude Rengerink K, Wiersma IC, Donker ME, Mol BW, Pajkrt E. Techniques for wound closure at caesarean section: a randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2012 Nov;165(1):47-52. doi: 10.1016/j.ejogrb.2012.07.019. Epub 2012 Aug 19. PMID 22910336
- [Background] Rousseau JA, Girard K, Turcot-Lemay L, Thomas N. A randomized study comparing skin closure in cesarean sections: staples vs subcuticular sutures. Am J Obstet Gynecol. 2009 Mar;200(3):265.e1-4. doi: 10.1016/j.ajog.2009.01.019. PMID 19254586
- [Background] Clay FS, Walsh CA, Walsh SR. Staples vs subcuticular sutures for skin closure at cesarean delivery: a metaanalysis of randomized controlled trials. Am J Obstet Gynecol. 2011 May;204(5):378-83. doi: 10.1016/j.ajog.2010.11.018. Epub 2010 Dec 31. PMID 21195384
- [Background] Tuuli MG, Rampersad RM, Carbone JF, Stamilio D, Macones GA, Odibo AO. Staples compared with subcuticular suture for skin closure after cesarean delivery: a systematic review and meta-analysis. Obstet Gynecol. 2011 Mar;117(3):682-690. doi: 10.1097/AOG.0b013e31820ad61e. PMID 21343772
- [Background] Mackeen AD, Berghella V, Larsen ML. Techniques and materials for skin closure in caesarean section. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD003577. doi: 10.1002/14651858.CD003577.pub3. PMID 23152219
- [Background] Shetty AA, Kumar VS, Morgan-Hough C, Georgeu GA, James KD, Nicholl JE. Comparing wound complication rates following closure of hip wounds with metallic skin staples or subcuticular vicryl suture: a prospective randomised trial. J Orthop Surg (Hong Kong). 2004 Dec;12(2):191-3. doi: 10.1177/230949900401200210. PMID 15621905
- [Background] Haymer DS, Marsh JL. Germ line and somatic instability of a white mutation in Drosophila mauritiana due to a transposable genetic element. Dev Genet. 1986;6(4):281-91. doi: 10.1002/dvg.1020060406. PMID 2840224
- [Background] Fick JL, Novo RE, Kirchhof N. Comparison of gross and histologic tissue responses of skin incisions closed by use of absorbable subcuticular staples, cutaneous metal staples, and polyglactin 910 suture in pigs. Am J Vet Res. 2005 Nov;66(11):1975-84. doi: 10.2460/ajvr.2005.66.1975. PMID 16334959
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752
- [Derived] Kuroki LM, Mullen MM, Massad LS, Wu N, Liu J, Mutch DG, Powell MA, Hagemann AR, Thaker PH, McCourt CK, Novetsky AP. Wound Complication Rates After Staples or Suture for Midline Vertical Skin Closure in Obese Women: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jul;130(1):91-99. doi: 10.1097/AOG.0000000000002061. PMID 28594761

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 173 participants were enrolled to the study but 8 participants had a change in their surgical procedure which deemed them ineligible for study enrollment and were excluded from the study before randomization to the arms.
Groups:
- 4-0 Monofilament Sutures: Skin closure using 4-0 monofilament sutures
Period: Overall Study
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Started | 85 | 80
Completed | 84 | 79
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures | Total
Number analyzed (Participants) | 84 | 79 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (13.2) | 57.1 (11.2) | 57.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 79 | 163
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 19 | 35
  White | 68 | 60 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 84 | 79 | 163
Body mass index (BMI) [Count of Participants; unit: Participants]
  30-39.9 | 60 | 49 | 109
  40-49.9 | 19 | 24 | 43
  50 or greater | 5 | 6 | 11
Prior Abdominal Surgery [Count of Participants; unit: Participants] | 51 | 53 | 104
Tobacco Use [Count of Participants; unit: Participants]
  Never | 44 | 59 | 103
  Former | 33 | 15 | 48
  Current | 7 | 5 | 12
Diabetes mellitus [Count of Participants; unit: Participants] | 27 | 19 | 46
Cardiovascular disease [Count of Participants; unit: Participants] | 58 | 57 | 115
Pulmonary disease [Count of Participants; unit: Participants] | 20 | 27 | 47
Prior malignancy [Count of Participants; unit: Participants] | 7 | 8 | 15
American Society of Anesthesiologists (ASA) class [Count of Participants; unit: Participants] — ASA 1 - Normal healthy patient ASA 2 - A patient with mild systemic disease ASA 3 - A patient with severe systemic disease that is a constant threat to life ASA 4 - A moribund patient who is not expected to survive without the operation
  Participants
    1-2 | 39 | 47 | 86
    3-4 | 45 | 32 | 77
Indications for surgery [Count of Participants; unit: Participants]
  Uterine cancer | 24 | 23 | 47
  Ovarian/fallopian/peritoneal cancer | 24 | 21 | 45
  Benign | 22 | 27 | 49
  Other | 11 | 5 | 16
  Synchronous primary | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Disruption or Infection (Wound Complications) Occurring Within 4-8 Weeks of the Date of the Primary Surgery.
Time Frame: 4-8 weeks post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Number analyzed (Participants) | 84 | 79
Participants | 28 | 25

2. Secondary Outcome: Incidence of Wound Disruption
Time Frame: 4-8 weeks post-surgery
Population: -Data on incidence of wound disruption was not collected on 9 patients in the stainless steel staple arm and 9 patients in the 4-0 Monocryl suture arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Number analyzed (Participants) | 75 | 70
Participants | 21 | 13

3. Secondary Outcome: Incidence of Wound Infection
Description: Purulent drainage, cellulitis, abscess, or a wound that requires drainage, debridement or antibiotics associated with a clinical diagnosis of infection.
Time Frame: 4-8 weeks post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Number analyzed (Participants) | 84 | 79
Participants | 1 | 1

4. Secondary Outcome: Operative Time
Description: Time from skin incision to the end of skin closure
Time Frame: During surgery
Population: Data was not collected from 3 patients in the stainless steel staple arm and 1 patient in the 4-0 Monocryl suture arm
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Number analyzed (Participants) | 81 | 78
minutes | 3 [2 to 4] | 11 [9 to 15]

5. Secondary Outcome: Analog Pain Score on Postoperative Days 3-4
Description: The highest pain score as recorded by nursing staff at a minimum of every 8 hours between 72-96 hours postoperatively.
Time Frame: 3-4 days post-surgery
Population: Data was not collected from any patients for this outcome measure
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cosmesis Score as Measured by the Stony Brook Scar Evaluation Score
Description: * Ranges from 0 (worst) to 5 (best)
  * Sum of width, height, color, hatch, and overall appearance where a better outcome has a value of 5 and a worse outcome has a value of 0
Time Frame: 4-8 weeks post-operative
Population: -Data was not collected from 10 patients in the Stainless Steel Staple arm and 9 patients in the 4-0 Monocryl Suture arm
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Number analyzed (Participants) | 74 | 70
units on a scale | 4 [3 to 5] | 5 [4 to 5]

7. Secondary Outcome: Median Patient Satisfaction Score of Scar Appearance
Description: Patients will be asked to rate the general appearance, location and comfort of the scar. This was collected as a continuous variable. Patients were given a paper survey and asked to please draw a single slash across a provided line indicating how satisfied they were with the appearance of their scar. The beginning of the line was designated "very unsatisfied" or 0% and the end of the line was "very satisfied" or 100%.
Time Frame: 4-8 weeks post-operative
Population: -Data was not collected on 13 patients in the Stainless Steel Staple arm and 12 patients in the 4-0 Monocryl Suture arm
Measure: Median (Inter-Quartile Range); unit: Patient Satisfaction Score
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Number analyzed (Participants) | 71 | 67
Patient Satisfaction Score | 68 [49 to 83] | 77 [52 to 87]

ADVERSE EVENTS:
Arm/Group | Stainless Steel Staples | 4-0 Monofilament Sutures
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/79
Other Adverse Events (participants affected / at risk) | 0/84 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes